CLINICAL TRIAL: NCT04074980
Title: Post CE Study: Evaluation of the Accuracy of INR Results From Patients Taking Phenprocoumon as Anticoagulant When Measured Using the Lumiradx INR Test
Brief Title: Evaluation of the Accuracy of INR Results From Patients Taking Phenprocoumon as Anticoagulant When Measured Using the Lumiradx INR Test
Acronym: VKA GERMANY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00013
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Hemostatic Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venous only (Experimental): One venous whole blood draw will be performed into two anti-coagulated collection tubes
  Interventions: Diagnostic Test: Venous blood draw
- Fingerstick and Venous (Experimental): One finger-stick sample of capillary blood (~10µl/sample) from each subject, will be applied directly to a unique test strip for immediate measurement of INR on the LumiraDx Instrument. One further fingerstick sample is then obtained (~10µl/sample) from a separate finger for immediate measurement of INR on the Coaguchek PRO. From each patient, one venous whole blood draw will also be performed into two anti-coagulated collection tubes.
  Interventions: Diagnostic Test: Venous and Fingerstick blood draws

INTERVENTIONS:
Diagnostic Test: Venous and Fingerstick blood draws — Fingerstick sampling to collect blood from subjects Venepuncture to collect blood samples from subjects
  Other Names: Venous and capillary blood draws
  Arms: Fingerstick and Venous
Diagnostic Test: Venous blood draw — Venepuncture to collect blood samples from subjects
  Arms: Venous only

SUMMARY:
This study is to evaluate the INR levels in patients taking phenprocoumon using the LumiraDx Point of Care INR test and comparing the results to the laboratory reference method , the ACL Elite Pro. Comparison will also be made with the Roche Coaguchek point of care INR test (point of care reference method). Performance will be demonstrated across a subject population of adult males and females in receipt of Phenprocoumon VKA therapy. This population is representative of the indications for use of the CE marked product. Operators will be trained clinical site staff. Venous plasma and capillary whole blood samples will be obtained from each subject in order to assess accuracy of the the LumiraDx Platform when compared to the reference devices (ACL Elite and Coaguchek Pro).

DETAILED DESCRIPTION:
Vitamin K antagonists (VKA) are a group of substances that reduce blood clotting by reducing the action of vitamin K. They are used in anticoagulant medications in the prevention of thrombosis. The drugs work by depleting the active form of the vitamin by inhibiting Vitamin K epoxide reductase and thus the recycling of inactive vitamin K back to the active reduced form. The most widely prescribed VKAs are Coumarins. This group is composed of several different structurally similar molecules and includes warfarin (Coumadin), acenocoumerol and phenprocoumon.

Within the EU there are country to country differences in preferential VKA prescription (1). In Germany and surrounding countries, Phenprocoumon (marketed as Marcoumar or Marcumar) is the most commonly prescribed. The majority of data supporting the development and validation of the LumriaDx INR test has used samples form patients taking Warfarin. The aim of this study is to evaluate the INR levels in patients taking phenprocoumon using the LumiraDx Point of Care INR test and comparing the results to the laboratory reference method , the ACL Elite Pro. Comparison will also be made with the Roche Coaguchek point of care INR test (point of care reference method).

This study is an observational, cross-sectional study with 100 patients in total. Devices used in this study are CE marked for INR measurement by healthcare professionals. This study will be conducted according to the principles of Good Clinical Practice (ICH GCP E6(R2)), International Conference on Harmonization Guidelines as applicable to devices, applicable geographical regulations and institutional research policies and procedures.

For part 1 of the study (25 patients), one venous whole blood draw will be performed (~9mL) into two anti-coagulated collection tubes (2 x 4.5mL 3.2% trisodium citrate). These tubes will then by processed to plasma by centrifugation, stored in Eppendorf tubes, labelled and frozen at -80ºC . These will then be transferred to the LumriaDx laboratory in Scotland, UK, for subsequent measurement of INR with the reference device IL ACL Elite Pro Coagulation Analyzer (ACL) and with the LumiraDx POC INR test.

For part 2 of the study (75 patients), one finger-stick sample of capillary blood (~10µl/sample) from each subject, will be applied directly to a unique test strip for immediate measurement of INR on the LumiraDx Instrument. One further fingerstick sample is then obtained (~10µl/sample) from a separate finger for immediate measurement of INR on the Coaguchek PRO. Post-testing, samples will be disposed securely. From each patient, one venous whole blood draw will also be performed (~9mL) into two anti-coagulated collection tubes (2 x 4.5mL 3.2% trisodium citrate). These tubes will then by processed to plasma by centrifugation, stored in Eppendorf tubes, labelled and frozen at -80ºC. These will then be transferred to the LumiraDx laboratory in Scotland, UK, for subsequent measurement of INR with the reference device IL ACL Elite Pro Coagulation Analyzer (ACL) and with the LumiraDx POC INR test.

INR results obtained will be used in comparative analyses of performance designed to meet the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Persons >18 years of age
* Willing and able to provide written informed consent and comply with study procedures
* Currently prescribed Phenprocoumon VKA Therapy
* Deemed medically appropriate for study participation by the Investigator

Exclusion Criteria:

* Subject has previously participated in this part of the study
* Subject is within 4 weeks of first prescription of Phenprocoumon
* Subject is taking a DOAC, or non-Phenprocoumon VKA therapy
* Confirmed or suspected pregnancy
* Vulnerable populations deemed inappropriate for study by the Investigator
* Deemed medically inappropriate for study by the Investigator (i.e. patients with a known inherited [e.g. haemophilia or von Willebrand's disease] or acquired [e.g. liver cirrhosis] condition likely to be associated with a coagulopathy; or patients receiving non-VKA anticoagulant medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
To determine the agreement of INR measurements of capillary whole blood as assessed by the LumiraDx POC INR test to INR measurements of venous plasma as assessed by the IL ACL ELITE PRO reference method. | 6 weeks
  Measurement of INR using Venous blood

SECONDARY OUTCOMES:
To determine the agreement of INR measurements of capillary whole blood as assessed by the LumiraDx POC INR test to INR measurements of capillary blood as assessed by Coaguchek Pro II. | 6 weeks
  Measurement of INR using Venous and capillary blood

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Voller, Principal Investigator — Haematologist
Locations (1):
- CLINICAL SITE Klinik am See, Rehabilitation Clinic for Cardiovascular Diseases, Ruedersdorf/Berlin., Rüdersdorf, Germany

IPD SHARING:
Plan to Share IPD: No